CLINICAL TRIAL: NCT07028905
Title: Clinical, Radiographical, and Histological Evaluation of Treatment Outcomes Following Different Caries Removal Strategies in Mature Permanent Teeth With Reversible Pulpitis (A Randomized Clinical Trial and Ex-vivo Study)
Brief Title: Deep Caries in Mature Teeth With Reversible Pulpitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Abeer mohamed shehata, Abeer Mohamed Shehata, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: deep caries in mature teeth
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Deep Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Total caries removal in primary caries (Active Comparator): Total caries removal Removal of all caries and application of bioactive material
  Interventions: Procedure: Total caries removal
- Total caries removal of secondary caries (Active Comparator): Total caries removal of caries of recurrent caries
  Interventions: Procedure: Total caries removal
- Partial caries removal of primary caries (Active Comparator): Partial caries removal and application of bioactive material
  Interventions: Procedure: Partial caries removal
- Partial caries removal of secondary caries (Active Comparator): Partical caries removal of recurrent caries
  Interventions: Procedure: Partial caries removal

INTERVENTIONS:
Procedure: Total caries removal — Total caries removal and application of bioactive material
  Other Names: Biodentin application
  Arms: Total caries removal in primary caries; Total caries removal of secondary caries
Procedure: Partial caries removal — Partial caries removal then application of biodentin
  Other Names: Biodentin
  Arms: Partial caries removal of primary caries; Partial caries removal of secondary caries

SUMMARY:
This clinical trial will be conducted to clinical, radiographical and histological evaluation of pulp condition with reversible pulpities after total and selective removal of primary and secondary caries (randomized clinical trial and exo-vivo study)

DETAILED DESCRIPTION:
Randomized clinical trial Sample size 144 case…

Randomization method used:

Sample size calculation was performed using R statistical analysis software version 4.3.2 for Windows

Outcome variables:

Pulp vitality and post operative pain Grouping classified into four groups as follows: The first group : total caries removal of primary caries(PTCR) 27 The second group: selective caries removal of primary caries(PSCR) The third group: total caries removal of secondary caries(STCR) The fourth group : selecive caries removal of secondary caries(SSCR)

Expected Time table:

2 years Recall of patient after 3,6,9 and 12 months 6 months for writing and 6 months for data analyzed

ELIGIBILITY:
Inclusion Criteria:

1. The patient's age from 18 years to 40 years old
2. Non -contributory medical history (ASA1)
3. Mature permanent posterior teeth with primary or secondary deep caries extending ≥ 2/3 of dentin
4. The tooth should give a positive response to cold testing
5. Clinical diagnosis of reversible pulpitis
6. The tooth is restorable via direct restoration, probing pocket depth and mobility are within normal limits
7. No signs of pulpal necrosis including sinus tract or swelling
8. No radiographic evidence of periapical changes indicative of apical periodontitis

Exclusion Criteria:

* Systemic medical conditions, pregnancy, alcoholic and smoker patients. 2- Teeth with spontaneous pain or percussion sensitivity in periodontal lesions, external or internal root resorption, sinus opening, mobility, or abscessed tooth. 3- Radiographic evidence of widened periodontal space, broken or interrupted lamina dura, and periapical radiolucency. 4- Intensified erosion damage or periodontitis. Patient reported clenching or bruxism, hopeless or non-restorable teeth. Immature teeth. 5- Patients with physical disabilities preventing tooth brushing. Patient had removable partial denture abutments, dental abscesses, pulp lesions, atypical facial pain, or pulpitis. 6- Patients had non-carious lesions like abrasion, erosion, attrition, or abfraction.

  7- Patients with history of antibiotic or analgesics intake within few days of operative intervention. 8- Patients with previously root canal-treated teeth. 9- Periodontally compromised teeth. 10-Teeth that will be extracted for periodontal or orthodontic reasons as it will conduct for histological evaluation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation ………. Radiographic evaluation: | 1year
  clinical evaluation: absence of pain , pulp vitality,
  ………. Radiographic evaluation: absence of any periapical lesion or recurrent caries

SECONDARY OUTCOMES:
histological evaluation and follow up | 1 year
  histological evaluation after one year. T (Time): follow up evaluation periods of pulp condition immediately post operative (base line ), after 3, 6, 9 and 12 month and exo-vivo study.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Mohmaed Shehata, Master, Principal Investigator — Minia University; Rasha Saad, lecturer, Study Director — Minia University; Mohammed Torky, Associate professor, Study Director — Minia University; Nermin Mahmoud, Associate professor, Study Director — Minia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taha NA, Ali MM, Abidin IZ, Khader YS. Pulp survival and postoperative treatment needs following selective vs. total caries removal in mature permanent teeth with reversible pulpitis: A randomized clinical trial. J Dent. 2024 Dec;151:105408. doi: 10.1016/j.jdent.2024.105408. Epub 2024 Oct 22. PMID 39442480
- [Background] Ahlawat M, Grewal MS, Goel M, Bhullar HK, Saurabh, Nagpal R. Direct Pulp Capping with Mineral Trioxide Aggregate and Biodentine in Cariously Exposed Molar Teeth: 1-Year Follow-up - An In vivo Study. J Pharm Bioallied Sci. 2022 Jul;14(Suppl 1):S983-S985. doi: 10.4103/jpbs.jpbs_837_21. Epub 2022 Jul 13. PMID 36110733
- [Background] Drouri S, El Merini H, Sy A, Jabri M. Evaluation of Direct and Indirect Pulp Capping With Biodentine in Vital Permanent Teeth With Deep Caries Lesions. Cureus. 2023 May 23;15(5):e39374. doi: 10.7759/cureus.39374. eCollection 2023 May. PMID 37250608